CLINICAL TRIAL: NCT05610930
Title: Effect of a New Graphically Modified Nutri-Score on the Objective Understanding of Foods' Nutritional Quality and Ultra-processing - a Randomised Controlled Trial
Brief Title: Is a Front-of-package Label Contaning Information on Both Nutrient Profile and Ultra-processing Well Understood?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Paris 13 (Other)
Responsible Party: Principal Investigator, Bernard Srour, Epidemiologist, University of Paris 13
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UParis13-BS
Record Dates: First submitted 2022-10-28; First posted 2022-11-09 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Objective Understanding of Nutritional Label

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): Participants received a questionnaire including 3 sets of images of food packaging, (brand blinded), categorized by food groups: 8 cookies, 7 breakfast cereals, and 7 ready-to-eat meals, but without front-of-pack nutritional label (in case the original Nutri-Score was displayed on the product, it was hidden by the investigators). They had the possibility to check the back-of-pack nutrition facts and ingredient information. First, they were asked which product they would intend to purchase in each category, and which product they thought to be the "healthiest". Then, participants were asked 1) to rank them according to their nutritional quality by identifying the first, the second and the third products with the best nutritional quality (in this order) and 2) to identify those that were ultra-processed.
- Experimental arm (Experimental): Participants received a questionnaire including 3 sets of images of real food product packaging (brand blinded), categorized by food groups: 8 cookies, 7 breakfast cereals, and 7 ready-to-eat meals, with the Nutri-Score 2.0 displayed on the front-of-pack of each product. First, they were asked which product they would intend to purchase in each category, and which product they thought to be the "healthiest". Then, participants were asked 1) to rank them according to their nutritional quality by identifying the first, the second and the third products with the best nutritional quality (in this order) and 2) to identify those that were ultra-processed. Last, a series of questions evaluated how participants of this arm perceived the Nutri-Score 2.0 and whether they found it helpful.
  Interventions: Other: Front-of-pack label NutriScore 2.0

INTERVENTIONS:
Other: Front-of-pack label NutriScore 2.0 — Participants in the experimental arm can see, in case the product is ultra-processed, a black banner surrounding the Nutri-Score, with the word "ultra-transformé", meaning ultra-processed, and no black banner otherwise. Participants in the control arm had no label at all. The intervention (the Nutri-Score 2.0) was added on the packaging on the products included in the 3 sets of images that participants recieved via the questionnaire.
  Arms: Experimental arm

SUMMARY:
A modified version of the Nutri-Score (Nutri-Score 2.0), containing an additional graphic mention when the product is ultra-processed, has been proposed. The investigators aim to study, in a randomised controlled trial design nested in the NutriNet-Santé cohort, the impact of this modified version on the objective understanding of foods' nutritional quality, and on the identification of UPFs as primary outcomes. They also aim to study as secondary outcomes the impact of this label on purchasing intentions and the product perceived as the healthiest.

DETAILED DESCRIPTION:
Two arms will be enrolled. The control arm will not have access to any FOP Label (the current situation in Europe), and the experimental arm will have access to Nutri-Score 2.0. Participants of both arms wil be asked to rank food products of 3 categories (breakfast cereals, cookies, ready-to-eat meals) according to their nutrient profile, and to identify ultra-processed foods.

ELIGIBILITY:
Inclusion Criteria:

Enrolled in the NutriNet-Santé cohort

Exclusion Criteria:

None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21159 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Objective understanding the nutritional quality. | Between 30 minutes and 1 hour (the time needed to fill the questionnaire)
  The answers of the participants on the corresponding questionnaire (via the NutriNet-Santé website) were expected to match the order according to which Nutri-Score ranks the 3 products (highest nutritional quality, second highest, third highest). In case of ex-æquos (i.e., two products having the same Nutri-Score), both were considered correct. Therefore, the number of correct answers for the nutritional dimension could range between 0 (no correct answers) to 9 (3 best products*3 food categories, all correct answers).
Objective understanding the ultra-processing dimension. | Between 30 minutes and 1 hour (the time needed to fill the questionnaire)
  Participants were expected to identify all UPFs on the corresponding questionnaire (via the NutriNet-Santé website). For each product, the answer was considered correct if an UPF was identified as such by the participant (the gold standard being the presence of the black banner of the Nutri-Score 2.0, corresponding to the NOVA 4 "ultra-processed" definition), and a non-UPF was identified as such. Therefore, the number of correct answers for the food processing dimension could range between 0 (no correct answers) and 22 (correct answer for all 22 products).

SECONDARY OUTCOMES:
Purchasing intentions | Between 30 minutes and 1 hour (the time needed to fill the questionnaire)
  Assessed with the question (in the corresponding questionnaire via the NutriNet-Santé website) : "Which of these products would you purchase more frequently?". This aimed to explore whether Nutri-Score 2.0 (the intervention) had an effect on the purchasing intentions.
Product perceived as the healthiest | Between 30 minutes and 1 hour (the time needed to fill the questionnaire)
  Assessed with the question (in the corresponding questionnaire via the NutriNet-Santé website) : "Which product seems the healthiest to you?". This aimed to explore whether Nutri-Score 2.0 (the intervention) had an effect on the product that the participants considered as the healthiest.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Srour, PhD, PharmD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Equipe de recherche en Epidémiologie nutritionnelle, Bobigny, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Srour B, Hercberg S, Galan P, Monteiro CA, Szabo de Edelenyi F, Bourhis L, Fialon M, Sarda B, Druesne-Pecollo N, Esseddik Y, Deschasaux-Tanguy M, Julia C, Touvier M. Effect of a new graphically modified Nutri-Score on the objective understanding of foods' nutrient profile and ultraprocessing: a randomised controlled trial. BMJ Nutr Prev Health. 2023 Jun;6(1):108-118. doi: 10.1136/bmjnph-2022-000599. Epub 2023 Jun 8. PMID 37484539